CLINICAL TRIAL: NCT05248113
Title: Intraoperative Electrically-evoked ABRs in Patients Undergoing Vestibular Schwannoma Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Harrison W Lin, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017-3885
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Deafness
Keywords: vestibular schwannoma; cochlear nerve; auditory prosthesis
MeSH Terms: conditions — Deafness; Neuroma, Acoustic

STUDY DESIGN:
Intervention Model Description: Test of feasibility of electrical stimulation of the cochlear nerve with a conventional bipolar nerve stimulator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intraoperative electrical stimulation of cochlear nerve (Experimental): Electrical stimulation of the cochlear nerve will be tested intraoperatively in patients undergoing vestibular schwannoma resection.
  Interventions: Device: Electrical stimulation of cochlear nerve

INTERVENTIONS:
Device: Electrical stimulation of cochlear nerve — Intraoperative electrical stimulation of the cochlear nerve in patients undergoing surgery for resection of vestibular schwannoma. Activation of the auditory system monitored with scalp recording of auditory brainstem response.

SUMMARY:
This is a study of the feasibility of activating the auditory system by an electrode in direct contact with the cochlear nerve.

DETAILED DESCRIPTION:
This is a feasibility study being conducted prior to development of a penetrating cochlear nerve stimulating electrode. Experiments will be conducted in patients who are undergoing surgery for resection of a vestibular schwannoma (VS). In the normal course of such a surgical procedure, the cochlear nerve is exposed and, in many cases, the cochlear nerve is resected or function of the cochlear nerve is otherwise disrupted. Typically, recording electrodes are placed on the scalp for the purpose of recording sound-evoked auditory brainstem responses (ABRs), which serve as a measure of the functional status of the cochlear nerve. In this intraoperative experimental procedure, a conventional bipolar nerve stimulating electrode will be placed in contact with the cochlear nerve and the nerve will be stimulated with electrical pulses. Activation of the auditory system by the electrical pulses will be evaluated by measurement of electrically-evoked ABRs, using the same scalp electrodes that are typically used for measurement of sound-evoked ABRs. The cochlear-nerve stimulating electrode will be in place only during the actual intraoperative test. No device will remain in the patient. The intraoperative experimental procedure is not intended to as a therapeutic measure for the patient's VS.

ELIGIBILITY:
Inclusion Criteria:

* Adults with the diagnosis of unilateral or bilateral vestibular schwannoma proven on radiographic imaging.
* Only patients with little or no hearing ability undergoing surgical resection of the tumor will be enrolled.

Exclusion Criteria:

* Women who are pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Auditory brainstem response | Recorded immediately during ongoing cochlear-nerve stimulation
  Electrical potentials recorded with scalp electrodes in response to electrical stimulation of the cochlear nerve

CONTACTS AND LOCATIONS:
Overall Officials: Harrison M Lin, MD, Principal Investigator — University of California, Irvine; John C Middlebrooks, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- UC Irvine Health, Pavilion II, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No